CLINICAL TRIAL: NCT02112344
Title: A Phase I Study of Intensity-modulated Radiotherapy in Patients With Squamous Cell Carcinoma of Unknown Primary (SCCUP) of the Head and Neck
Brief Title: A Study of Intensity-modulated Radiotherapy in Patients With Squamous Cell Carcinoma of Unknown Primary (SCCUP) of the Head and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 2823
Record Dates: First submitted 2014-03-13; First posted 2014-04-11 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total mucosal irradiation (Experimental)
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT

SUMMARY:
Squamous cell carcinoma of unknown primary (SCCUP) site metastatic to cervical lymph nodes at presentation is a relatively rare entity forming about 2% of all head and neck carcinomas.

Typically patients are treated with ipsilateral modified radical neck dissection (MRND) and post-operative radiotherapy (PORT) or chemoradiotherapy.

There is a lack of consensus on the radiotherapy target volumes that should be treated after neck dissection. The most common radiotherapy techniques are either unilateral cervical lymph node irradiation to achieve local control in the ipsilateral neck or TMI of the head and neck region with the aim of eradicating the primary and the microscopic neck disease.

Treatment of the ipsilateral hemi-neck alone is of low toxicity and may achieve local control in the cervical nodes. Potential occult primary sites in the head and neck mucosa, and any sub-clinical metastatic disease in the contralateral side of the neck are left untreated. If a primary tumour subsequently becomes apparent the previous radiotherapy may make further radiotherapy difficult to deliver.

Some groups recommend bilateral neck and total mucosal irradiation in this setting claiming improved local control. With conventional radiotherapy technique this is at the price of significant acute toxicity and chronic morbidity, mainly xerostomia with its associated complications and effects on quality of life (QOL).

Intensity modulated radiotherapy (IMRT) has been shown to reduce the dose to salivary gland tissue and consequently may reduce the incidence of xerostomia and improve quality of life (QOL) in head and neck cancer patients.

An analysis of parotid-sparing IMRT at the University of Michigan established a mean dose threshold for both stimulated (26 Gy), and unstimulated (24 Gy) saliva flow rates. For the same end-point (less than 25% of flow at baseline one year post radiation) Roesink et al established a TD50 of 39 Gy.

The investigators performed a planning study to assess the feasibility of IMRT to spare the parotid gland while delivering bilateral neck and TMI. The mean dose to the contralateral parotid gland using IMRT was below the threshold of 24 Gy for unstimulated salivary flow, predicting a fairly low risk of radiation induced xerostomia. The mean dose to the ipsilateral parotid gland was 32 Gy which was below the TD50 dose based on the Roesink data.

This study assesses the safety and tolerability of delivering IMRT in clinical practice to treat patients with SCCUP of the head and neck region, who require bilateral neck and pan-mucosal irradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinomas metastatic to cervical lymph node with occult primary requiring bilateral neck and pan mucosal irradiation.
2. Radiotherapy either as primary therapy or post-operative (adjuvant irradiation).
3. Neoadjuvant and concomitant chemotherapy are permitted.
4. All patients must be suitable to attend regular follow-up and undergo toxicity assessment.
5. Stage T0, N1-3, M0 disease
6. WHO Performance Status 0-1.
7. Patient should have a negative PET/CT scan for a primary tumour.

Exclusion Criteria:

1. Previous radiotherapy to the head and neck region
2. Previous malignancy except non-melanoma skin cancer
3. Previous or concurrent illness which in the investigators opinion would interfere with either completion of therapy or follow-up
4. Prophylactic use of amifostine or pilocarpine is not allowed
5. Brachytherapy is not allowed as part of the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-07; Primary Completion 2010-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of delivering IMRT | 7 weeks after starting radiotherapy
  Feasibility of delivering IMRT in this setting i.e. all the patients completing the radiotherapy protocol without treatment breaks due to toxicity.

SECONDARY OUTCOMES:
Incidence of acute dermatitis | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of >grade 1 late xerostomia | 5 years
  Outcome measured at 3, 6, 12, 18, 24 months after RT.
Number of patients who do not relapse at the local site | 5 years
  Local control assessed at 3, 6 months, then every 6 months to 5 years.
Overall survival | 5 years
  Assessed at 3 and 6 months then every 6 months to 5 years.
Incidence of acute alopecia | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of >grade 1 acute dysphagia | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of > grade 1 acute mucositis | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of acute radiation induced pain | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of >grade 1 acute xerostomia | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of acute radiation induced fatigue | 3 months after RT
  Outcome measured at baseline, weeks 1-6 during RT. Weeks 1-4 and 8 after RT.
Incidence of > grade 1 late dysphagia | 5 years after RT
  Outcome measured at 3, 6, 12, 18, 24 months after RT.
Incidence of late oesophageal stricture | 5 years after RT
  Outcome measured at 3, 6, 12, 18, 24 months after RT.
Incidence of >grade 1 late hoarse voice | 5 years after RT
  Outcome measured at 3, 6, 12, 18, 24 months after RT.
Incidence of late radiation induced neurological dysfunction | 5 years
  Outcome measured at 3, 6, 12, 18, 24 months after RT.
Incidence of >grade1 late skin toxicity | 5 years after RT
  Outcome measured at 3, 6, 12, 18, 24 months after RT.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Nutting, PhD, Principal Investigator — Royal Marsden NHS Foundation Trust